CLINICAL TRIAL: NCT06377241
Title: A Proof-of-concept Pilot Study to Determine the Efficacy of SensifyAware and Retinal Imaging in Differentiating Mild Cognitive Impairment (MCI) From Cognitively Unimpaired Controls (HC)
Brief Title: ScentAware and OCT in MCI vs HC
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1436; A536000 (Other: UW Madison); SMPH/OPHTHAL&VIS SCI/GEN (Other: UW Madison); Protocol Version 9/20/2024 (Other: UW Madison)
Record Dates: First submitted 2024-04-03; First posted 2024-04-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: No cognitive impairment, and no family history of Alzheimer's disease
  Interventions: Device: ScentAware; Device: UPSIT
- Cohort 2: No cognitive impairment, with a family history of Alzheimer's disease
  Interventions: Device: ScentAware; Device: UPSIT
- Cohort 3: Mild cognitive impairment due to Alzheimer's disease
  Interventions: Device: ScentAware; Device: UPSIT

INTERVENTIONS:
Device: ScentAware — ScentAware is a smell test
Device: UPSIT — UPSIT is a smell test

SUMMARY:
The goal of this clinical trial is to learn whether a new smell test works as well as the standard clinical smell test, if there is a link between sense of smell and variations in the retina, and if these results could be used as a way to identify early stages of Alzheimer's disease. The main questions it aims to answer are:

* Whether the test is as effective and reliable as the standard test
* Whether there is a link between the results of the smell test and the structure of the back of the eye

Participants will:

* complete a short questionnaire
* have pictures of the inside of their eyes taken
* perform two smell tests

ELIGIBILITY:
Inclusion Criteria:

* Adults who are ≥ 50 and ≤ 80 years of age
* Fluent in English
* Able to provide written consent
* Able to complete a 2.5-3-hour clinical visit, including sitting for spectral domain optical coherence tomography (SD-OCT) imaging for 30 minutes and taking cognitive and olfactory tests for 90-120 minutes
* Cognitive Ability and Family History of Alzheimer's Disease/Mild Cognitive Impairment (AD/MCI):

  * Cohort 1: Cognitively unimpaired, no family history of MCI or AD, and MMSE ≥ 26
  * Cohort 2: Cognitively unimpaired, a positive family history of MCI or AD, and MMSE ≥ 26
  * Cohort 3: An MMSE score > 22 and ≤ 25 and either

    * Clinically diagnosed MCI due to AD
    * A participant in a Wisconsin ADRC research registry with either clinically diagnosed MCI or self-reported MCI
* Cohorts 1 and 2: proficient in independent use of mobile smart devices

Exclusion Criteria:

* A history of significant ocular or nasal trauma that required medical/surgical intervention
* A history of intraocular surgery except cataract extraction
* A cataract extraction within 3 months prior to enrollment
* Diagnosis of visually significant intraocular disease (such as late-stage age-related macular degeneration, glaucoma, or other optic nerve conditions related to brain tumor or multiple sclerosis), drug related vision loss or retinal damage
* Optic neuritis on both eyes
* Current use of medications that may interfere with olfactory functions
* Current use of hydroxychloroquine and tamoxifen, which are known to cause retinal toxicity that may confound OCT interpretation
* A history of recurrent or chronic oto-pharyngeal-laryngeal (ORL) disease (such as chronic rhinitis, nasal polyposis, or sinus disease), head trauma, toxic exposures, upper respiratory infections at time of assessment
* A family history or diagnosis of other neurodegenerative diseases (e.g., multiple sclerosis, Parkinson's disease, Huntington's disease) or conditions that, in the opinion of the Investigators, may affect cognitive or olfactory functions
* Olfactory loss due to COVID (current olfactory loss and/or temporary loss that has been regained)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (50-80 years of age) in three cohorts:
  Cohort 1: 10 participants cognitively unimpaired with no family history of AD Cohort 2: 10 participants cognitively unimpaired with a family history of AD Cohort 3: 10 participants with clinically diagnosed MCI or from the Wisconsin ADRC registry and clinically diagnosed or self-reported MCI
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Compare test scores of ScentAware olfactory test to the scores of the University of Pennsylvania Smell Identification Test (UPSIT) olfactory test in a clinical setting | Baseline
  Performance of ScentAware and UPSIT odor identification score will be performed using Receiver Operating Characteristic (ROC) Curve analysis. Area under the ROC curve (AUC) will be used to determine diagnostic accuracy. An AUC ranges from 0 to 1. Higher AUC values indicate better sensitivity.
Compare ScentAware test results conducted with support from clinical staff to the test results when ScentAware test was self-administered independently | One month post baseline
  Performance of ScentAware and UPSIT odor identification score will be performed using Receiver Operating Characteristic (ROC) Curve analysis. Area under the ROC curve (AUC) will be used to determine diagnostic accuracy. An AUC ranges from 0 to 1. Higher AUC values indicate better sensitivity.
Compare UPSIT test results conducted with support from clinical staff to the test results when ScentAware test was self-administered independently | One month post baseline
  Performance of ScentAware and UPSIT odor identification score will be performed using Receiver Operating Characteristic (ROC) Curve analysis. Area under the ROC curve (AUC) will be used to determine diagnostic accuracy. An AUC ranges from 0 to 1. Higher AUC values indicate better sensitivity.

SECONDARY OUTCOMES:
Compare baseline ScentAware test scores between cohorts | Baseline
Compare baseline UPSIT test scores between cohorts | Baseline
Compare baseline ScentAware test scores to the retinal nerve fiber layer (RNFL) thickness | Baseline
Compare baseline UPSIT test scores to the retinal nerve fiber layer (RNFL) thickness | Baseline
Compare baseline ScentAware test scores to the ganglion cell layer (GCL) thickness | Baseline
Compare baseline UPSIT test scores to the ganglion cell layer (GCL) thickness | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sanbrita Mondal, OD, Principal Investigator — University of Wisconsin, Madison; Kathleen Schildroth, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States